CLINICAL TRIAL: NCT03095053
Title: PGT for Aneuploidy Does Not Enhance Live Birth in Young Patients (≤35 Years): a Randomized Controlled Trial of Single Blastocyst Frozen Embryo Transfers (ClinicalTrials.Gov ID: NCT03095053)
Brief Title: PGT-A Versus Blastocyst Morphology Selection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya IVF (Other)
Responsible Party: Principal Investigator, Kevin Coetzee, Scientific advisor, Antalya IVF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: euploid versus morphology; Optimizing implantation in FET (Other: Antalya IVF)
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Pregnancy
Keywords: morphological score; preimplantation genetic testing; frozen embryo transfer; blastocyst

STUDY DESIGN:
Intervention Model Description: single-centre randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGT-A group (Active Comparator): Next Generation sequencing preimplantation genetic testing for aneuploidy
  Interventions: Procedure: comprehensive chromosome screening
- Morphology group (No Intervention): morphological assessment of blastocyst by light microscope

INTERVENTIONS:
Procedure: comprehensive chromosome screening — Biopsy Blastocysts with morphological grades of ≥2BB will be biopsied on day 5 of in vitro embryo culture. Biopsies will be performed using a Hamilton Thorne Zilos laser (Hamilton Thorne, MA, USA), with 3-10 trophectoderm cells removed from the blastocysts.
  Comprehensive chromosome screening All trophectoderm biopsies will be processed for analysis by Next-Generation Sequencing (NGS, Illumina, California, USA).
  Arms: PGT-A group

SUMMARY:
Introduction Embryo aneuploidy is likely the leading cause of implantation failure in IVF cycles. Since the inception of IVF, non-invasive morphology based scoring has been the most widely used embryo selection method, resulting in relatively low embryo implantation rates. Our understanding of the optimal conditions required for in vitro embryo culture in IVF has advanced significantly over the past two decades. The implementation of improved in vitro embryo culture technologies (i.e., culture media and incubators) has resulted in an increase in the number of good quality embryos and consequently in increased numbers of blastocysts. While blastocyst transfers have seemingly improved the reproductive outcomes of IVF, they still remain suboptimal. The main objective of this randomized controlled trial (RCT) will be to investigate whether preimplantation genetic testing (i.e., PGT with comprehensive chromosome screening (CCS)) for aneuploidy is a superior embryo selection method, with the live birth outcomes of euploid blastocyst frozen embryo transfers (FET) compared with the LB outcomes of unknown-ploidy blastocyst FET, with blastocysts selected on (standard) morphological score.

Methods This RCT will be conducted at a single private IVF centre performing routine segmented-IVF, with intracytoplasmic sperm injection (ICSI), blastocyst freeze-all, and artificial frozen embryo transfer (art-FET). Normo-ovulatory infertile patients, with maternal age ≤35 years and at least two blastocysts with a morphology score of 2BB cryopreserved, will be randomized by computer-generated randomized allocation to either the PGT or morphology arm of the trial. All transfers will be single embryo transfers (SET), with only the first FET cycles following freeze-all to be analyzed.

Consent and Ethics Akdeniz University Medical Faculty Clinical Research Ethics Committee has approved the trial (reference number: 2015/399), with anonymized results to be released in ClinicalTrials.gov. All patients will provide informed consent, which included an agreement for the use of anonymised data for research and SET.

DETAILED DESCRIPTION:
Introduction Embryo aneuploidy is likely the leading cause of implantation failure in IVF cycles. Since the inception of IVF, non-invasive morphology based scoring has been the most widely used embryo selection method, resulting in relatively low embryo implantation rates. Embryo morphology assessment methods have significant limitations (i.e., the assessments are subjective and the method uses fixed time-point assessments to define dynamic embryo development) and shortcomings (i.e., exposes embryos to sub-optimal conditions during assessment). Notwithstanding the limitations and shortcomings of this method its use worldwide has continued, because it is a relatively simple and non-invasive method and its scores have been shown to be (moderately) positively correlated to embryo euploidy, ongoing pregnancy, and live birth (Van Royen et al., 1999, Ahlstrom et al., 2011, Forman et al., 2013, Capalbo et al., 2014, Oron et al., 2014, Rhenman et al., 2015).

However multiple gestations still represents one of the most significant complications in IVF, which are mainly the result of multiple-embryo embryo transfers, with multiple-embryo transfers used to overcome the relatively low embryo implantation rates in IVF. Our understanding of the optimal conditions required for in vitro embryo culture in IVF has advanced significantly in the past two decades. The implementation of improved in vitro embryo culture technologies (i.e., culture media and incubators) has resulted in an increase in the number of good quality embryos and consequently in the numbers of blastocysts. While blastocyst transfers have seemingly improved the reproductive outcomes in IVF, the use of SET and PGT technologies have revealed embryo implantation still to be sub-optimal (Schoolcraft et al., 2013). New CCS platforms are a major breakthrough in PGT, allowing 24-chromosome screening to be performed with high degree of accuracy from single cells (Harper and Harton, 2010). The evidence that morphology scores were only moderately associated with euploidy and that the transfer of PGT predicted euploid embryos resulted in higher implantation rates (Dahdouh et al., 2015), has seen the continued use of morphology-based scoring methods increasingly being challenged.

In addition to all the other advances in IVF, significant improvements have also been made in cryopreservation technologies. These improvements have resulted in significant improvements in frozen-thawed embryo survival (i.e. minimizing of risks), post-thaw developmental competence (Cobo et al., 2012; Balaban et al., 2008), and in the reproductive outcomes of FET (Evans et al., 2014; Ozgur et al., 2015). The benefits of FET include; the transfer of embryos to a more physiologic endometrium (i.e., early luteal phase), the ability to time transfers more accurately, and the ability to use patient-specific endometrial preparations (Casper and Yanushpolsky, 2016, Franasiak et al., 2016; Groenewoud et al., 2013, Yarali et al., 2016).

Moreover, the hypotheses of PGT requires to be confirmed in further robust RCT before its implementation in routine IVF.

Objectives The primary objective of this RCT will be to investigate whether PGT for aneuploidy as a blastocyst selection method is superior to standard morphology scoring blastocyst selection, comparing the reproductive outcomes in FET cycles. The decision to transfer all blastocysts in FET will eliminate any potential impact of ovarian stimulation confounding on endometrial receptivity and to use freeze-all cycles will allow the use of the primary blastocysts of blastocyst cohorts. The primary outcome measure of this trial will be LB, with a LB defined as a pregnancy cycle delivering at >20 weeks of gestation.

Secondary objectives The secondary objective of the RCT will be to investigate whether euploid blastocyst transfer results in reduced miscarriage, with a miscarriage defined as a clinical pregnancy lost at <20 weeks of gestation.

Keywords: blastocyst; comprehensive chromosome screening; euploidy; frozen embryo transfer

ELIGIBILITY:
Inclusion Criteria:

Patient-couples eligible for inclusion in the trial must satisfy the following criteria; female age of ≤35 years, female body mass index (BMI) of ≥18 or ≤35 kg/m2, antral follicle count (AFC) of ≥10, normo-ovulatory, intend to use autologous oocytes, and have ≥2 blastocysts with a morphological score of 2BB on day 5 of embryo development

Exclusion Criteria:

Patient couples will be excluded from the trial for the following reasons, patients with drug contraindications, patients with pathophysiology unrelated to reproduction, patients with intrauterine pathophysiologies, patients with no blastocysts, patients with <2 blastocysts with a morphological score of 2BB.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 302 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Coetzee, PhD, Principal Investigator — Antalya IVF
Locations (1):
- Antalya IVF, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahlstrom A, Westin C, Reismer E, Wikland M, Hardarson T. Trophectoderm morphology: an important parameter for predicting live birth after single blastocyst transfer. Hum Reprod. 2011 Dec;26(12):3289-96. doi: 10.1093/humrep/der325. Epub 2011 Oct 3. PMID 21972253
- [Result] Balaban B, Urman B, Ata B, Isiklar A, Larman MG, Hamilton R, Gardner DK. A randomized controlled study of human Day 3 embryo cryopreservation by slow freezing or vitrification: vitrification is associated with higher survival, metabolism and blastocyst formation. Hum Reprod. 2008 Sep;23(9):1976-82. doi: 10.1093/humrep/den222. Epub 2008 Jun 10. PMID 18544577
- [Result] Capalbo A, Rienzi L, Cimadomo D, Maggiulli R, Elliott T, Wright G, Nagy ZP, Ubaldi FM. Correlation between standard blastocyst morphology, euploidy and implantation: an observational study in two centers involving 956 screened blastocysts. Hum Reprod. 2014 Jun;29(6):1173-81. doi: 10.1093/humrep/deu033. Epub 2014 Feb 26. PMID 24578475
- [Result] Casper RF, Yanushpolsky EH. Optimal endometrial preparation for frozen embryo transfer cycles: window of implantation and progesterone support. Fertil Steril. 2016 Apr;105(4):867-72. doi: 10.1016/j.fertnstert.2016.01.006. Epub 2016 Jan 25. PMID 26820769
- [Result] Cobo A, de los Santos MJ, Castello D, Gamiz P, Campos P, Remohi J. Outcomes of vitrified early cleavage-stage and blastocyst-stage embryos in a cryopreservation program: evaluation of 3,150 warming cycles. Fertil Steril. 2012 Nov;98(5):1138-46.e1. doi: 10.1016/j.fertnstert.2012.07.1107. Epub 2012 Aug 3. PMID 22862909
- [Result] Dahdouh EM, Balayla J, Garcia-Velasco JA. Comprehensive chromosome screening improves embryo selection: a meta-analysis. Fertil Steril. 2015 Dec;104(6):1503-12. doi: 10.1016/j.fertnstert.2015.08.038. Epub 2015 Sep 16. PMID 26385405
- [Result] Evans J, Hannan NJ, Edgell TA, Vollenhoven BJ, Lutjen PJ, Osianlis T, Salamonsen LA, Rombauts LJ. Fresh versus frozen embryo transfer: backing clinical decisions with scientific and clinical evidence. Hum Reprod Update. 2014 Nov-Dec;20(6):808-21. doi: 10.1093/humupd/dmu027. Epub 2014 Jun 10. PMID 24916455
- [Result] Forman EJ, Upham KM, Cheng M, Zhao T, Hong KH, Treff NR, Scott RT Jr. Comprehensive chromosome screening alters traditional morphology-based embryo selection: a prospective study of 100 consecutive cycles of planned fresh euploid blastocyst transfer. Fertil Steril. 2013 Sep;100(3):718-24. doi: 10.1016/j.fertnstert.2013.04.043. Epub 2013 May 30. PMID 23725804
- [Result] Franasiak JM, Ruiz-Alonso M, Scott RT, Simon C. Both slowly developing embryos and a variable pace of luteal endometrial progression may conspire to prevent normal birth in spite of a capable embryo. Fertil Steril. 2016 Apr;105(4):861-6. doi: 10.1016/j.fertnstert.2016.02.030. PMID 26940791
- [Result] Groenewoud ER, Cantineau AE, Kollen BJ, Macklon NS, Cohlen BJ. What is the optimal means of preparing the endometrium in frozen-thawed embryo transfer cycles? A systematic review and meta-analysis. Hum Reprod Update. 2013 Sep-Oct;19(5):458-70. doi: 10.1093/humupd/dmt030. Epub 2013 Jul 2. PMID 23820515
- [Result] Harper JC, Harton G. The use of arrays in preimplantation genetic diagnosis and screening. Fertil Steril. 2010 Sep;94(4):1173-1177. doi: 10.1016/j.fertnstert.2010.04.064. Epub 2010 Jun 25. PMID 20579641
- [Result] Oron G, Son WY, Buckett W, Tulandi T, Holzer H. The association between embryo quality and perinatal outcome of singletons born after single embryo transfers: a pilot study. Hum Reprod. 2014 Jul;29(7):1444-51. doi: 10.1093/humrep/deu079. Epub 2014 May 8. PMID 24812313
- [Result] Ozgur K, Berkkanoglu M, Bulut H, Isikli A, Coetzee K. Higher clinical pregnancy rates from frozen-thawed blastocyst transfers compared to fresh blastocyst transfers: a retrospective matched-cohort study. J Assist Reprod Genet. 2015 Oct;32(10):1483-90. doi: 10.1007/s10815-015-0576-1. Epub 2015 Sep 23. PMID 26400506
- [Result] Rhenman A, Berglund L, Brodin T, Olovsson M, Milton K, Hadziosmanovic N, Holte J. Which set of embryo variables is most predictive for live birth? A prospective study in 6252 single embryo transfers to construct an embryo score for the ranking and selection of embryos. Hum Reprod. 2015 Jan;30(1):28-36. doi: 10.1093/humrep/deu295. Epub 2014 Nov 5. PMID 25376459
- [Result] Schoolcraft WB, Katz-Jaffe MG. Comprehensive chromosome screening of trophectoderm with vitrification facilitates elective single-embryo transfer for infertile women with advanced maternal age. Fertil Steril. 2013 Sep;100(3):615-9. doi: 10.1016/j.fertnstert.2013.07.1972. PMID 23993664
- [Result] Van Royen E, Mangelschots K, De Neubourg D, Valkenburg M, Van de Meerssche M, Ryckaert G, Eestermans W, Gerris J. Characterization of a top quality embryo, a step towards single-embryo transfer. Hum Reprod. 1999 Sep;14(9):2345-9. doi: 10.1093/humrep/14.9.2345. PMID 10469708
- [Result] Yarali H, Polat M, Mumusoglu S, Yarali I, Bozdag G. Preparation of endometrium for frozen embryo replacement cycles: a systematic review and meta-analysis. J Assist Reprod Genet. 2016 Oct;33(10):1287-1304. doi: 10.1007/s10815-016-0787-0. Epub 2016 Aug 22. PMID 27549760
- [Derived] Ozgur K, Berkkanoglu M, Bulut H, Yoruk GDA, Candurmaz NN, Coetzee K. Single best euploid versus single best unknown-ploidy blastocyst frozen embryo transfers: a randomized controlled trial. J Assist Reprod Genet. 2019 Apr;36(4):629-636. doi: 10.1007/s10815-018-01399-1. Epub 2019 Jan 7. PMID 30617927

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patient population of the RCT consisted of patients who underwent autologous blastocyst freeze-all IVF cycles between March and October 2016, at a private IVF center
Pre-assignment Details: Excluded (N =82) Patients with no blastocyst Patients with <2 blastocysts Patients with only one 2BB blastocyst
Groups:
- PGT-A Group: comprehensive chromosome screening
  comprehensive chromosome screening: Biopsy Blastocysts with morphological grades of ≥2BB will be biopsied on day 5 of in vitro embryo culture. Biopsies will be performed using a Hamilton Thorne Zilos laser (Hamilton Thorne, MA, USA), with 3-10 trophectoderm cells removed from the blastocysts.
  Comprehensive chromosome screening All trophectoderm biopsies will be processed for analysis by Next-Generation Sequencing (NGS, Illumina, California, USA).
Period: Overall Study
Arm/Group | PGT-A Group | Morphology Group
Started | 109 (All blastocysts scored morphologically PGT-A of the single best blastocyst from the cohort) | 111 (All blastocysts scored morphologically)
Completed | 80 (29 excluded as blastocyst was predicted to be aneuploid) | 111
Not Completed | 29 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PGT-A Group | Morphology Group | Total
Number analyzed (Participants) | 109 | 111 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] — Female patients aged >18 and ≤35 years
  years | 28.5 (3.71) | 28.3 (3.24) | 28.4 (3.48)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Infertile couples included based on female factors
  Participants | 109 | 111 | 220
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Mean (Standard Deviation); unit: kg/m^2"] — Body mass index (BMI) is quantitative classification of weight using the measures of height and weight
  kg/m^2" | 25.3 (4.11) | 25.1 (4.49) | 25.2 (4.3)
Antral follicle count [Mean (Standard Deviation); unit: number of antral follicles] — transvaginal ultrasound examination
  number of antral follicles | 21.9 (14.16) | 24.2 (16.28) | 23.1 (15.27)
Infertility duration [Mean (Standard Deviation); unit: years] — years of unprotected sex without successful pregnancy
  years | 3.9 (2.64) | 4.4 (3.10) | 4.2 (2.89)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With a Live Birth
Description: A live birth cycle was defined as a cycle with a delivery after 20 weeks of gestation.
Time Frame: >20 weeks gestation
Population: The live birth rates in the study trial groups
Measure: Count of Participants; unit: Participants
Groups:
- Euploid Subgroup: comprehensive chromosome screening
  comprehensive chromosome screening: Biopsy Blastocysts with morphological grades of ≥2BB will be biopsied on day 5 of in vitro embryo culture. Biopsies will be performed using a Hamilton Thorne Zilos laser (Hamilton Thorne, MA, USA), with 3-10 trophectoderm cells removed from the blastocysts.
  Comprehensive chromosome screening All trophectoderm biopsies will be processed for analysis by Next-Generation Sequencing (NGS, Illumina, California, USA).
Arm/Group | Euploid Subgroup | Morphology Group
Number analyzed (Participants) | 80 | 111
Participants | 45 | 65

2. Secondary Outcome: The Percentage of Patients With a Clinical Pregnancy
Description: A clinical pregnancy was defined as a cycle with a fetal sac observed on ultrasound after 5 weeks of gestation
Time Frame: >5 weeks of gestation
Population: The clinical pregnancy rates in the study trial groups
Measure: Count of Participants; unit: Participants
Arm/Group | Euploid Subgroup | Morphology Group
Number analyzed (Participants) | 80 | 111
Participants | 49 | 76

3. Secondary Outcome: The Percentage of Pregnancies That Miscarried
Description: A miscarriage was defined as the loss of a clinical pregnancy before 20 weeks of gestation.
Time Frame: <20 weeks
Population: The miscarriage rates in the study trial groups
Measure: Count of Participants; unit: Participants
Arm/Group | Euploid Subgroup | Morphology Group
Number analyzed (Participants) | 49 | 76
Participants | 3 | 11

ADVERSE EVENTS:
Time Frame: Patients were followed-up for adverse events from the start date of ovarian stimulation to the final outcome of segmented IVF treatment; approximately 37 weeks for not pregnant patients and 77 weeks for pregnant patients
Arm/Group | PGT-A Group | Morphology Group
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/111
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/111
Other Adverse Events (participants affected / at risk) | 0/109 | 0/111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT03095053/Prot_SAP_000.pdf